CLINICAL TRIAL: NCT03108547
Title: Hair Cortisol and Testosterone Levels in Patients With Sarcoidosis Associated Fatigue
Brief Title: Hair Cortisol and Testosterone Levels in Patients With Sarcoidosis
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Marlies Wijsenbeek, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2014-206
Record Dates: First submitted 2017-03-31; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; Scalp hair cortisol and testosterone; Fatigue; Biomarker; Psychological distress
MeSH Terms: conditions — Sarcoidosis; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Scalp hair string
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Sarcoidosis - fatigued: Men and women with sarcoidosis and a score of ≥ 22 on the Fatigue Assessment Scale. A small hair sample will be cut and the participants will be asked to complete questionnaires on fatigue, anxiety, depression, stress and quality of life.
  Interventions: Other: Determination of scalp hair steroids
- Sarcoidosis - non-fatigued: Men and women with sarcoidosis and a score of < 22 on the Fatigue Assessment Scale. A small hair sample will be cut and the participants will be asked to complete questionnaires on fatigue, anxiety, depression, stress and quality of life.
  Interventions: Other: Determination of scalp hair steroids
- Healthy controls: Hair steroid values of a previously collected normal values study in adults will be used as healthy controls
  Interventions: Other: Determination of scalp hair steroids

INTERVENTIONS:
Other: Determination of scalp hair steroids

SUMMARY:
The investigators studied whether scalp hair cortisol and testosterone levels differed between sarcoidosis patients both with and without fatigue and healthy controls.

DETAILED DESCRIPTION:
Rationale: Fatigue is a common symptom in patients with sarcoidosis and has great impact on quality of life. Several aspects in the pathogenesis of sarcoidosis and co-morbidities accompanying sarcoidosis could contribute to fatigue. However, until now the etiology of fatigue in sarcoidosis is unknown. Measurements of steroid hormones in scalp hair could possibly be directional in elucidating the underlying mechanism and could also be used as a screening and follow up tool in interventional studies.

Objective: A pilot to investigate whether cortisol and testosterone levels measured in hair differ between patients with sarcoidosis related fatigue, sarcoidosis patients without fatigue and healthy subjects.

Study design: A prospective observational study, using hair samples of sarcoidosis patients with and without fatigue, compared to an already existing age matched healthy control group.

Study population: Adult sarcoidosis patients at the outpatient clinic of the pulmonary department of the Erasmus MC, Rotterdam Main study parameters/endpoints: Cortisol and testosterone levels in scalp hair, correlation with Fatigue Assessment Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Diagnosis of sarcoidosis based on consistent clinical features/BAL fluid analysis/ PA according to the latest ATS/ERS/WASOG statement on sarcoidosis
* Able to speak, read and write in Dutch
* Presence of sarcoidosis related fatigue, defined as a ≥ 22 score on the Fatigue Assessment Scale
* Other causes of fatigue are excluded or contributing comorbidities are optimally treated (e.g. OSAS, hypothyroidism or anemia)

Exclusion Criteria:

* Unable to understand questionnaires (intellectual impaired or language barrier)
* Hair length < 1 cm
* Use of systemic and/ or inhalation steroids in the last year
* Use of methylphenidate (Ritalin) < 1 month before the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Diagnosis of sarcoidosis based on consistent clinical features/BAL fluid analysis/ PA according to the latest ATS/ERS/WASOG statement on sarcoidosis
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-06-13 (Actual); Primary Completion 2015-01-05 (Actual); Study Completion 2015-01-05 (Actual)

PRIMARY OUTCOMES:
Scalp hair cortisol differences between sarcoidosis patients with and without fatigue and healthy controls | 1 month
  Differences between patients with sarcoidosis related fatigue, sarcoidosis patients without fatigue, and healthy controls

SECONDARY OUTCOMES:
Scalp hair testosterone differences between sarcoidosis patients with and without fatigue and healthy controls | 1 month
  Differences between patients with sarcoidosis related fatigue, sarcoidosis patients without fatigue, and healthy controls
Scalp hair cortisone differences between sarcoidosis patients with and without fatigue and healthy controls | 1 month
  Differences between patients with sarcoidosis related fatigue, sarcoidosis patients without fatigue, and healthy controls
Fatigue Assessment Scale (FAS) | 1 day
  A short validated questionnaire to assess fatigue in sarcoidosis, and its relation to scalp hair steroids
King's Sarcoidosis Questionnaire (KSQ) | 1 day
  A validated questionnaire to assess sarcoidosis-related health status, and its relation to scalp hair steroids
EuroQol-5D-5L (EQ-5D-5L) | 1 day
  A validated generic questionnaire to assess general health status, and its relation to scalp hair steroids
Short Form-36 (SF-36) | 1 day
  A validated generic questionnaire to assess health-related quality of life, and its relation to scalp hair steroids
Perceived Stress Scale | 1 day
  A validated questionnaire to assess perception of stress, and its relation to scalp hair steroids
Hospital Anxiety and Depression Scale | 1 day
  A validated questionnaire to identify presence of depression and anxiety, and their relation to scalp hair steroids
% predicted forced vital capacity (FVC) | 1 day
  To assess the relationship between scalp hair steroids and FVC
% predicted diffusion capacity of carbon monoxide (DLCO) | 1 day
  To assess the relationship between scalp hair steroids and DLCO
6-minute walk distance test (6MWT) | 1 day
  To assess the relationship between scalp hair steroids and 6MWT
Waist circumference | 1 day
  To assess the relationship between scalp hair steroids and waist circumference
Body Mass Index (BMI) | 1 day
  To assess the relationship between scalp hair steroids and BMI

CONTACTS AND LOCATIONS:
Overall Officials: M. S. Wijsenbeek, MD, PhD, Principal Investigator — Erasmus University Medical Center, Rotterdam, the Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Manen MJG, Wester VL, van Rossum EFC, van den Toorn LM, Dorst KY, de Rijke YB, Wijsenbeek MS. Scalp hair cortisol and testosterone levels in patients with sarcoidosis. PLoS One. 2019 Jun 14;14(6):e0215763. doi: 10.1371/journal.pone.0215763. eCollection 2019. PMID 31199799